CLINICAL TRIAL: NCT00461071
Title: RCT on the Use of Psychoeducation for Bulimia Nervosa in Young Women
Brief Title: Randomised Controlled Study on the Use of Psychoeducation for Bulimia Nervosa in Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: National Bank of Austria (Other Government)
Responsible Party: Principal Investigator, Dr. Andreas Karwautz, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AP11957ONB
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Bulimia Nervosa
Keywords: Bulimia nervosa; Guided Self-help; Psycho-education
MeSH Terms: conditions — Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Internet-based self-help (Active Comparator): Internet-based self-help behavioural
  Interventions: Behavioral: Guided Self-help for Bulimia nervosa
- Bibliotherapy (Active Comparator): bibliotherapy
  Interventions: Behavioral: Guided Self-help for Bulimia nervosa

INTERVENTIONS:
Behavioral: Guided Self-help for Bulimia nervosa — bibliotherapy

SUMMARY:
The purpose of this study is to evaluate the effectivity of guided self-help via Internet and bibliotherapy in the treatment of bulimia nervosa (BN) in young women.

DETAILED DESCRIPTION:
Eating disorders and especially bulimia nervosa are psychiatric diseases, affecting 2-4% of women. An intervention such as guided self-help via manuals (bibliotherapy) is a well accepted approach and accepted. Development of new technologies in recent years allows delivery of psychotherapy via CD-ROMs and web-based interfaces. These new technologies have not yet been implemented in Austria in treating bulimia nervosa (BN) patients. In particular patients will be involved, who would not attend medical care regularly. The aim of our study is therefore to deliver guided self-help via an internet platform (supported by email contacts) for 100 patients with BN and to investigate the practicability and effectivity of this approach as well as compliance of patients in this group.

Patients will be found and contacted via internet, get specialized medical investigations, medical care and support via emails. As control group 100 patients with bulimia are treated with bibliotherapy only. Beside effectivity, predictors of outcome (clinical, comorbidity, indication to change, personality) are investigated.

The proposed study is a randomised controlled trial for effectivity and practicability of new technologies in psychiatric treatment research.

This is not a psychotherapy study but a study on psychoeducation, an approach which offers new and helpful opportunities for this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bulimia nervosa purging-type
* BMI > 18 or age corresponding BMI in patients younger than 18y.
* Access to Internet available

Exclusion Criteria:

* Severe depression, alcohol- or drug abuse
* acute suicidality

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2007-04; Primary Completion 2008-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Eating disorder symptomatology after 3 months and after 7 months | december 2009
  Eating disorder symptomatology after 3 months and after 7 months

SECONDARY OUTCOMES:
Predictors for best outcome | december 2009
  Predictors for best outcome
motivation for change | dec 2009
  motivation for change

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karwautz, MD, Prof, Study Director — Medical University of Vienna, Dep. of Children and Adolescent Psychiatry
Locations (1):
- Medical University of Vienna, Dep. of Children and Adolescent Psychiatry, Vienna, Austria

REFERENCES:
- [Derived] Wagner G, Penelo E, Nobis G, Mayrhofer A, Wanner C, Schau J, Spitzer M, Gwinner P, Trofaier ML, Imgart H, Fernandez-Aranda F, Karwautz A. Predictors for good therapeutic outcome and drop-out in technology assisted guided self-help in the treatment of bulimia nervosa and bulimia like phenotype. Eur Eat Disord Rev. 2015 Mar;23(2):163-9. doi: 10.1002/erv.2336. Epub 2014 Dec 1. PMID 25448409
- [Derived] Wagner G, Wagner G, Penelo E, Nobis G, Mayerhofer A, Schau J, Spitzer M, Imgart H, Karwautz A. Is technology assisted guided self-help successful in treating female adolescents with bulimia nervosa? Neuropsychiatr. 2013;27(2):66-73. doi: 10.1007/s40211-013-0062-x. Epub 2013 Apr 23. PMID 23609487
- [Derived] Wagner G, Penelo E, Wanner C, Gwinner P, Trofaier ML, Imgart H, Waldherr K, Wober-Bingol C, Karwautz AF. Internet-delivered cognitive-behavioural therapy v. conventional guided self-help for bulimia nervosa: long-term evaluation of a randomised controlled trial. Br J Psychiatry. 2013 Feb;202:135-41. doi: 10.1192/bjp.bp.111.098582. Epub 2012 Dec 6. PMID 23222037
- See also: related Information — http://www.ess-stoerung.eu